CLINICAL TRIAL: NCT01158261
Title: A Prospective, Single-Arm, Observational, Non-interventional Study for EVICEL ™ Fibrin Sealant (Human) When Used as an Adjunct to Haemostasis in Vascular Surgery
Brief Title: The Evicel Post-Authorization Surveillance Study
Status: Completed | Type: Observational
Sponsor: Ethicon, Inc. (Industry)
Collaborators: OMRIX Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 400-08-004
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-07

CONDITIONS: Peripheral Vascular Disease; Hemorrhage
Keywords: hemostasis
MeSH Terms: conditions — Peripheral Vascular Diseases; Hemorrhage | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vascular Surgery Subjects Treated with EVICEL
  Interventions: Biological: EVICEL ™ Fibrin Sealant (Human)

INTERVENTIONS:
Biological: EVICEL ™ Fibrin Sealant (Human) — Commercial Evicel
  Other Names: Fibrin Sealant (Human)

SUMMARY:
The objective of this non-interventional Post Authorisation Safety Surveillance (PASS) study is to observe the clinical safety performance of EVICEL when used as suture support for haemostasis in vascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, 18 years or older, requiring elective, primary or repeat vascular procedures with at least one end-to-side anastomosis to the femoral artery or to an upper extremity artery
* EVICEL Fibrin Sealant is used as an adjunct to obtain haemostasis at a target anastomosis/es
* Subjects must be willing to and capable of participating in the study, and provide written informed consent

Exclusion Criteria:

* Subjects with known intolerance to blood products
* Subjects unwilling to receive blood products
* Subjects with any intra-operative findings that may preclude the use of a fibrin sealant to control suture line anastomotic bleeding
* Subject participating in another study with an investigational (pre-approved) drug or device within 30 days of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects requiring elective vascular procedures
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-06; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kocharian, MD, Study Director — Ethicon, Inc.
Locations (2):
- United States (2):
  - Baptist Health Medical Center, Jacksonville, Florida
  - Memorial Hospital, Jacksonville, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled 04 June 2010 and the last subject was enrolled 15 April 2014. The last data point collected for the trial was 21 May 2014.
Groups:
- EVICEL® Fibrin Sealant (Human): All procedures were performed according to the surgeon's standard of care. EVICEL® Fibrin Sealant was prepared and used according to the current approved instructions for use and product indication. The anastomoses were constructed and checked for bleeding. Anastomotic repair sutures were placed and then, if bleeding requiring adjunctive treatment persisted, arterial clamps were re-applied. The surgeon then applied EVICEL® by dripping onto the anastomotic site/s according to his/her standard practice. Arterial clamps were removed approximately 1-minute following the end of product application to allow for curing. All subjects were followed for approximately 4 weeks following surgery.
Period: Overall Study
Arm/Group | EVICEL® Fibrin Sealant (Human)
Started | 300
Completed | 283
Not Completed | 17
Not completed — Lost to Follow-up | 9
Not completed — Death | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | EVICEL® Fibrin Sealant (Human)
Number analyzed (Participants) | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 151
  >=65 years | 149
Age, Continuous [Median (Full Range); unit: years] — The study population has a mean age of 62.2 years (std 13.9). The median is reported in the table below.
  years | 64 [19 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 180
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 105
  White | 185
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 300
BMI (grouped) [Number; unit: participants]
  Underweight | 5
  Normal | 84
  Overweight | 79
  Obese | 108
  Morbidly obese | 24
History of Smoking [Number; unit: participants]
  Never smoked | 108
  Ex-smoker | 136
  Current smoker | 56

OUTCOME MEASURES:

1. Primary Outcome: Specific Safety Parameters
Description: * Incidence of graft occlusion
  * Incidence of adverse events potentially related to non-graft thrombotic events
  * Incidence of bleeding events
Time Frame: Up to 4-weeks post-operatively
Population: From participant flow, 283 subjects completed the study; One subject lost to follow-up had 4-week information in hospital records.
Measure: Number; unit: participants
Arm/Group | EVICEL® Fibrin Sealant (Human)
Number analyzed (Participants) | 284
participants
  Graft Occlusion | 12
  AE potentially related to non-graft thrombosis | 7
  Bleeding events | 0

ADVERSE EVENTS:
Time Frame: From enrollment through the 4-week follow-up
Groups:
- EVICEL® Fibrin Sealant (Human): An adverse event (AE) was defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of the EVICEL® product. For the purpose of this protocol, an AE was any untoward medical occurrence in a study subject that may be related or possibly related to the EVICEL® product. The relatedness to EVICEL® was based on the investigator's assessment.
  In the original version of the protocol, the SAE definition did not require that the AE be related or possibly related to the treatment. This discrepancy with the AE definition resulted in the sites reporting non-EVICEL® related AEs and SAEs prior to the amended protocol implementation.
Arm/Group | EVICEL® Fibrin Sealant (Human)
Serious Adverse Events (participants affected / at risk) | 22/300
Other Adverse Events (participants affected / at risk) | 23/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EVICEL® Fibrin Sealant (Human) (N=300)
Angina pectoris (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Groin abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Ateriovenous fistula site complication (Injury, poisoning and procedural complications) | 2
Eschar (Injury, poisoning and procedural complications) | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 2
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
Steal syndrome (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EVICEL® Fibrin Sealant (Human) (N=300)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 4
Vascular graft occlusion (Injury, poisoning and procedural complications) | 3
Hypotension (Vascular disorders) | 2
Steal Syndrome (Vascular disorders) | 2
Nodal rhythm (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Graft infection (Infections and infestations) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1
Urine analysis abnormal (Investigations) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Urethral stenosis (Renal and urinary disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Limitations of the study include the small number of centers involved and the observational nature of the design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No